CLINICAL TRIAL: NCT05700253
Title: Comparing Pain Outcomes of Cooled Radiofrequency Ablation and Hyaluronic Acid Therapies for Chronic Osteoarthritis Knee Patients
Brief Title: Comparing Pain Outcomes of Treatment Strategies for Osteoarthritis Knee Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Prit Anand Singh, Senior Consultant, Department of Anaesthesia and Surgical Intensive Care, Changi General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Osteoarthritis01
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis, Knee; Pain
Keywords: cooled radiofrequency ablation; hyaluronic acid injection
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooled Radiofrequency Ablation (Experimental): Relieves pain by blocking pain signals via the deactivation of nerve structures using radiofrequency energy.
  Interventions: Device: Cooled Radiofrequency Ablation
- Hyaluronic Acid Injection (Active Comparator): Injection of hyaluronic acid into the affected knee provides lubrication and shock absorption.
  Interventions: Device: Hyaluronic Acid Injection

INTERVENTIONS:
Device: Cooled Radiofrequency Ablation — Image-guided genicular nerve ablation will be performed with the Coolief System (COOLIEF* CRFA; Avanos Medical).
  Arms: Cooled Radiofrequency Ablation
Device: Hyaluronic Acid Injection — Synvisc-One ([Hylan G-F 20]; Sanofi) will be administered as a single intra-articular dose (6 mL).
  Arms: Hyaluronic Acid Injection

SUMMARY:
The goal of this clinical trial is to compare two different pain relief techniques (cooled radiofrequency ablation (CRFA) and hyaluronic acid (HA) injection) for patients with knee osteoarthritis (OA) over a period of 6 months. The main questions it aims to answer are:

* the extent of reduction of pain score and the proportion of subjects ("responders") whose knee pain is reduced by at least 50% from baseline up to 6 months after treatment in the two treatment groups.
* the safety of the two treatment modalities.

Participants will undergo a nerve block test to determine if they would experience pain relief from blocking of nerve signals. Responders will be randomised to receive one of the two treatments for their knee pain. Researchers will compare the pain intensity of CRFA and HA injection groups at baseline, 2 weeks, 1 month, 3 months and 6 months post-treatment using validated questionnaires.

DETAILED DESCRIPTION:
This study will be a single-centred, open-label, prospective randomized controlled study to compare the extent of OA-related knee pain relief between subjects who undergo radiofrequency lesioning (COOLIEF* CRFA; Avanos Medical) of the genicular nerves and subjects who receive a single intra-articular HA injection (Synvisc-One [Hylan G-F 20]; Sanofi). Study subjects will receive CRFA or HA injection in a 1:1 randomization scheme, with post-treatment data collection at 2 weeks, 1 month, 3 months and 6 months. Six months was chosen as the duration of follow-up as that is the expected duration of medical improvement following HA injection for chronic knee pain. Knee pain, function, overall subject impressions of treatment, quality of life, pain medication use, and adverse events will be compared among the treatment cohorts. The study is open-label as blinding is not possible due to the differences in administration of injection and CRFA, hence both the patient and the investigator will be aware of the treatment type.

The primary endpoints will be the extent of reduction of pain score measured via 11-point visual analogue scale (VAS). Secondary outcomes will include proportion of subjects ("responders") whose knee pain is reduced by at least 50% from baseline up to 6 months after treatment, patients' overall knee pain score as measured via Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), subjects' perception of treatment effect as measured via Knee injury and Osteoarthritis Outcome Score (KOOS), patients' perception of treatment effect via Global Perceived Effect (GPE) score and health related quality of life via EuroQol-5 Dimensions 5 Level (EQ-5D-5L). Assessments of these study endpoints will be made at baseline, 2 weeks, 1 month, 3 months and 6 months following treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Able to understand the informed consent form and provide written informed consent and able to complete outcome measures
3. Chronic knee pain for longer than 3 months that interferes with functional activities (for example, ambulation, prolonged standing, etc.)
4. Continued pain in the target knee despite at least 3 months of conservative treatments, including activity modification, home exercise, protective weight bearing, and/or analgesics (for example, acetaminophen or non-steroidal anti-inflammatory drugs [NSAIDs] etc.)
5. Positive response (defined as a decrease in numeric pain scores of at least 50%) to a single genicular nerve block of the index knee
6. Pain on VAS ≥ 6 on an 11-point scale for the index knee
7. Radiologic confirmation of arthritis (x-ray/MRI/CT) of OA grade of 2 (mild), 3 (moderate) or 4 (severe) noted within 6 months for the index knee
8. An intra-articular HA injection is indicated as an appropriate treatment option
9. WOMAC Knee Score group at baseline of Score of ≥ 2 (0 to 4 scale) on WOMAC question 1 (Pain) and a mean score of ≥ 1.5 on all five questions of the WOMAC pain subscale
10. Agree to see one physician (study physician) for knee pain during the study period
11. Willing to delay any surgical intervention for the index knee for the period of the study follow up
12. Willing to comply with the requirements of this protocol for the full duration of the study

Exclusion Criteria:

1. Evidence of inflammatory arthritis (for example, rheumatoid arthritis) or other systemic inflammatory condition (for example, gout, fibromyalgia) that could cause knee pain
2. Evidence of neuropathic pain secondary to other causes (e.g., sciatica), apart from OA knee, affecting the index knee
3. Previous or pending lower limb amputation
4. Intra-articular steroid or PRP injection or Radiofrequency lesioning into the index knee within 180 days from randomization
5. Hyaluronic acid injection, PRP injection, stem cell, or arthroscopic debridement/lavage injection into the index knee within 180 days from randomization
6. Prior partial, resurfacing, or total knee arthroplasty of the index knee (residual hardware)
7. Clinically significant ligamentous laxity of the index knee
8. Clinically significant valgus/varus deformities or evidence of pathology (other than osteoarthritis of knee) that materially affects gait or function of the knee or is the underlying cause of the knee pain and/or functional limitations
9. Body mass index (BMI) > 45 kg/m2 or < 18 kg/m2
10. Extremely thin patients and those with minimal subcutaneous tissue thickness that would not accommodate a radiofrequency lesion of up to 14 mm in diameter to limit the risk of skin burns
11. Pending or active compensation claim, litigation, or disability remuneration (secondary gain)
12. Pregnant, nursing or intent of becoming pregnant during the study period
13. Chronic pain associated with significant psychosocial dysfunction
14. Patients with known psychiatric history including severe mental health issues.
15. Allergies to any of the medications to be used during the procedures, including known hypersensitivity (allergy) to hyaluronate preparations or allergies to avian or avian-derived products (including eggs, feathers, or poultry)
16. Active joint infection or systemic or localized infection at needle entry sites (subject may be considered for inclusion once infection is resolved)
17. History of uncontrolled coagulopathy, ongoing coagulation treatment that cannot be safely interrupted for procedure, or unexplained or uncontrollable bleeding that is not correctable
18. Identifiable anatomical variability that would materially alter the procedure as described in the protocol
19. Within the preceding 2 years, subject has suffered from active narcotic addiction, substance, or alcohol abuse
20. Current prescribed opioid medications greater than 60 milligrams morphine equivalent daily opioid dose
21. Uncontrolled immunosuppression (e.g., AIDS, cancer, diabetes, etc.)
22. Subject currently implanted with pacemaker, stimulator or defibrillator
23. Participating in another clinical trial/investigation within 30 days prior to signing informed consent
24. Subject unwilling or unable to comply with follow up schedule or protocol requirements

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Extent of reduction of pain score | 6 months
  11-point Visual Analogue Scale

SECONDARY OUTCOMES:
Proportion of subjects ("responders") whose knee pain is reduced by at least 50% from baseline up to 6 months after treatment. | 6 months
  11-point Visual Analogue Scale
Overall knee pain score | 6 months
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Opinion of knee injury and treatment outcomes | 6 months
  Knee injury and Osteoarthritis Outcome Score (KOOS)
Perception of treatment effect | 6 months
  Global Perceived Effect (GPE) score
Health related quality of life | 6 months
  EuroQol-5 Dimensions 5 Level (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Prit Anand Singh, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu L, Li Y, Si H, Zeng Y, Li M, Liu Y, Shen B. Radiofrequency Ablation in Cooled Monopolar or Conventional Bipolar Modality Yields More Beneficial Short-Term Clinical Outcomes Versus Other Treatments for Knee Osteoarthritis: A Systematic Review and Network Meta-Analysis of Randomized Controlled Trials. Arthroscopy. 2022 Jul;38(7):2287-2302. doi: 10.1016/j.arthro.2022.01.048. Epub 2022 Feb 12. PMID 35157969
- [Background] Oladeji LO, Cook JL. Cooled Radio Frequency Ablation for the Treatment of Osteoarthritis-Related Knee Pain: Evidence, Indications, and Outcomes. J Knee Surg. 2019 Jan;32(1):65-71. doi: 10.1055/s-0038-1675418. Epub 2018 Nov 5. PMID 30396206
- [Background] Chen AF, Khalouf F, Zora K, DePalma M, Kohan L, Guirguis M, Beall D, Loudermilk E, Pingree MJ, Badiola I, Lyman J. Cooled radiofrequency ablation provides extended clinical utility in the management of knee osteoarthritis: 12-month results from a prospective, multi-center, randomized, cross-over trial comparing cooled radiofrequency ablation to a single hyaluronic acid injection. BMC Musculoskelet Disord. 2020 Jun 9;21(1):363. doi: 10.1186/s12891-020-03380-5. PMID 32517739
- [Background] Chen AF, Khalouf F, Zora K, DePalma M, Kohan L, Guirguis M, Beall D, Loudermilk E, Pingree M, Badiola I, Lyman J. Cooled Radiofrequency Ablation Compared with a Single Injection of Hyaluronic Acid for Chronic Knee Pain: A Multicenter, Randomized Clinical Trial Demonstrating Greater Efficacy and Equivalent Safety for Cooled Radiofrequency Ablation. J Bone Joint Surg Am. 2020 Sep 2;102(17):1501-1510. doi: 10.2106/JBJS.19.00935. PMID 32898379
- [Background] Lyman J, Khalouf F, Zora K, DePalma M, Loudermilk E, Guiguis M, Beall D, Kohan L, Chen AF. Cooled radiofrequency ablation of genicular nerves provides 24-Month durability in the management of osteoarthritic knee pain: Outcomes from a prospective, multicenter, randomized trial. Pain Pract. 2022 Jul;22(6):571-581. doi: 10.1111/papr.13139. Epub 2022 Jun 29. PMID 35716058
- See also: Avanos Coolief System — https://avanospainmanagement.com/solutions/chronic-pain/genicular-neurotomy/